CLINICAL TRIAL: NCT00683449
Title: A Phase II, Randomized, Modified Single-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety and Efficacy of MN-221 When Administered Intravenously as an Adjunct to Standard Therapy to Adults With an Acute Exacerbation of Asthma
Brief Title: Study Evaluating the Safety and Effects of MN-221 in Subjects Experiencing an Acute Exacerbation of Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data from Dose Groups 1,2 and other MN-221 studies resulted in the determination of a more appropriate dosing scheme for MN-221 in subjects with asthma.
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MN-221-CL-006
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Asthma; Status Asthmaticus
Keywords: Asthma; Dose-Escalation; Controlled; MN-221
MeSH Terms: conditions — Asthma; Status Asthmaticus | interventions — bedoradrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV infusion of MN-221 (Experimental): MN-221 total dose of 240 mcg
  Interventions: Drug: Dose Group 1; Drug: Dose Group 2; Drug: Dose Group 3
- MN-221 PLACEBO (Placebo Comparator): i.v. infusion of MN-221 Placebo for 15 min
  Interventions: Drug: MN-221 placebo

INTERVENTIONS:
Drug: Dose Group 1 — IV infusion of MN-221 16 mcg/min for 15 min; total dose of 240 mcg
  Other Names: bedoradrine
  Arms: IV infusion of MN-221
Drug: MN-221 placebo — i.v. infusion of placebo for 15 minutes
  Other Names: bedoradrine
  Arms: MN-221 PLACEBO
Drug: Dose Group 2 — i.v. infusion of MN-221 30 mcg/min for 15 minutes (total dose of 450 mcg)
  Other Names: bedoradrine
  Arms: IV infusion of MN-221
Drug: Dose Group 3 — i.v. infusion of MN-221 16 mcg/min for 15 minutes followed by 8 mcg/min for 105 minutes (total dose = 1,080 mcg)
  Other Names: bedoradrine
  Arms: IV infusion of MN-221

SUMMARY:
The objective of this clinical study is to examine the safety and effectiveness of intravenous MN-221 compared to placebo when administered as an adjunct to standard therapy in subjects experiencing an acute exacerbation of asthma.

DETAILED DESCRIPTION:
This is a randomized, modified single-blind, placebo-controlled dose escalation, multi-center Emergency Department (ED) study. Each subject will receive MN-221 or placebo administered through a continuous intravenous infusion in addition to the standardized care treatment for an acute exacerbation of asthma. The study is a modified single-blind design where the subject and the Investigator will be blinded.

Upon presentation to the ED for assessment and treatment for an acute exacerbation of asthma the subject should receive standardized care consistent with the National Asthma Education and Prevention Program (NAEPP) guidelines.

Once the subject has received the standardized initial treatment regimen and has been assessed for response to that treatment (signs and symptoms of acute asthma exacerbation), an informed consent to participate in the study will be obtained, study entry criteria will be reviewed, a 12-lead ECG will be performed, a dyspnea index scale assessment will be conducted, and spirometry will be performed. If the subject's FEV1 is ≤ 55% of predicted and the subject meets all other study entry criteria the subject will be randomized to receive either MN-221 or placebo. Throughout the screening process the subject will continue to receive the appropriate medical care consistent with the NAEPP guidelines for the treatment of acute exacerbations of asthma.

There will be up to three dose groups with generally twelve subjects in each group. Subjects enrolled in the study will receive an intravenous infusion of MN-221 study drug or placebo. Generally six subjects will be randomized to receive MN-221 and generally six subjects will be randomized to receive placebo in each dose group.

The initial dose group will be randomized to receive:

* 16 μg/min of MN-221 for 15 minutes (total dose of 240 μg) or placebo.

Subsequent dose groups will receive the following proposed doses:

* 30 μg/min for 15 minutes (total dose of 450 μg) or placebo, and
* 16 μg/min for 15 minutes followed by 8 μg/min for 105 minutes (total dose of 1,080 μg) or placebo.

During the study treatment period, the subject will continue to receive the following standard treatment and assessment until the subject's FEV1 reaches ≥ 70% of predicted:

* Assessment of subject's signs and symptoms;
* Complete a dyspnea index scale;
* Supplemental oxygen to maintain oxygen saturation as measured by pulse oximetry of ≥ 90%;
* Albuterol (2.5 mg) via nebulizer given hourly; NOTE: Albuterol (2.5 mg) via nebulizer may be given up to every 20 minutes if deemed to be indicated by the Investigator.
* Ipratropium (0.5 mg) via nebulizer may be given every hour if deemed to be indicated by the Investigator.
* Spirometry completed within 10 minutes of nebulizer treatments; followed by,
* Reassessment of signs and symptoms. If the subject does not improve to FEV1 ≥ 70% of predicted during the study treatment period, the subject may continue to receive further treatment including hospital admission at the discretion of the Investigator. The study will be approximately 6.5 hours in length (Hour -1.5 to Hour 5) while the subject remains in the ED. Safety, efficacy and PK parameters will be monitored throughout the treatment period. An initial 24-hour post-randomization follow-up visit will be completed to evaluate the subject's health status as well as for safety and PK parameters. A second follow-up contact will be completed by telephone seven days post-randomization for safety purposes and to evaluate the subject's health status.

A risk/benefit evaluation will be performed by the study's Safety Review Committee at each dose level. The occurrence of clinical signs, symptoms, laboratory abnormalities, ECG abnormalities suggesting toxicity, or results of efficacy analyses (FEV1, dyspnea index scale), may result in a decision to modify the proposed planned dose escalations, to repeat a dose level, or to not evaluate any additional dose(s) of MN-221.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. Have self-reported history of physician-diagnosed and treated asthma for ≥ 3 months;
3. Have a diagnosis of an acute exacerbation of asthma upon presentation at the ED as defined by dyspnea and evidence of bronchospasm in an individual with a known history of asthma;
4. Upon presentation to the ED the treatment provided included:

   * A brief history and physical examination that includes vital signs, auscultation, assessments of accessory respiratory muscle usage and the level of dyspnea the subject is experiencing;
   * Supplemental oxygen given to maintain oxygen saturation as measured by pulse oximetry of ≥ 90%;
   * Two doses of inhaled beta2-agonist (defined as albuterol 5 mg) via nebulizer (each dose given sequentially up to approximately every 20 minutes); simultaneously with
   * Two doses of an inhaled anti-cholinergic agent (defined as ipratropium 0.5 mg) via nebulizer (each dose given sequentially up to approximately every20 minutes);
   * One dose of corticosteroid of at least 60 mg given orally (prednisone) or intravenously (methylprednisolone); and
5. Have a FEV1 ≤ 55% within 10 minutes of completing the treatment described in Inclusion Criterion #4;
6. Have a negative urine pregnancy test if you are females of childbearing potential;
7. Have ECG with no dysrhythmias (except sinus tachycardia);
8. Have no clinical or electrocardiographic signs of ischemic heart disease as determined by the Investigator; and
9. Have signed the informed consent obtained prior to starting any study procedures.

Exclusion criteria:

1. Have a current or prior diagnosis or suspected diagnosis of COPD or other chronic lung disease other than asthma;
2. Have presence of pneumonia;
3. Have presence of significant other respiratory dysfunction such as pneumothorax, pneumomediastinum, or pulmonary edema;
4. Have known or suspected vocal cord dysfunction syndrome;
5. Have presence of aspirated foreign body (known or suspected);
6. Have a history or any current clinical evidence suggesting cardiomyopathy or congestive heart failure;
7. Have a history or presence of tachyarrhythmias, with the exception of sinus tachycardia;
8. Have a heart rate ≥ maximum heart rate: (maximum predicted HR [220-age]-30); OR Heart rate ≥ 150 bpm;
9. Have hypokalemia, defined as a potassium level ≤ 3.0 mg/dL according to the point-of-care device level obtained at Screening;
10. Have significant cardiac, renal, hepatic, endocrine, metabolic, neurologic or other systemic disease. A significant disease will be defined as one which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study or the subject's ability to participate in the trial;
11. Have a self-reported history of greater than 15 pack-yr smoking history;
12. Have a fever ≥ 101.5º F;
13. Have uncontrolled hypertension defined as a blood pressure ≥ 170/100 mm Hg;
14. Have the need for immediate intubation as determined by the Investigator;
15. Are a pregnant or lactating female;
16. Have participated in another clinical study with an investigational drug within 30 days of randomization;
17. Have a positive urine drug screen for cocaine, methamphetamine or PCP;
18. Have a known allergy to MN-221 or any of the other components of the MN-221 drug product ;
19. Have a known allergy to other beta agonists;
20. Have had previous exposure to MN-221; or
21. Have used of theophylline, beta blockers, diuretics, digoxin, MAO inhibitors, or tricyclic antidepressants within 2 weeks prior to randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kalafer, MD, Study Director — MediciNova
Locations (9):
- United States (9):
  - Maricopa Medical Center; Dept. of Emergency Medicine, Phoenix, Arizona
  - LAC + USC Medical Center, Los Angeles, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine; Div. of Emergency Medicine, St Louis, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lewis LM, Ferguson I, House SL, Aubuchon K, Schneider J, Johnson K, Matsuda K. Albuterol administration is commonly associated with increases in serum lactate in patients with asthma treated for acute exacerbation of asthma. Chest. 2014 Jan;145(1):53-59. doi: 10.1378/chest.13-0930. PMID 23949578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon presentation to the Emergency Department (ED) at a hospital participating in the study with an acute exacerbation of asthma, the Principal Investigator (ED physician) discussed the study with the potential subject.
Pre-assignment Details: Some subjects were consented for the study, but upon screening, failed to meet the inclusion and exclusion criteria, had an FEV1 > 50%, or refused to participate.
Groups:
- 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes: Initial dose: 16 μg/min of MN-221 for 15 minutes (total 240 μg). After safety data review meeting, chose escalation doses: 1) 30 μg/min for 15 minutes (total 450 μg), and 2) 16 μg/min for 15 minutes plus 8 μg/min for 105 minutes (total dose of 1,080 μg).Until the subject's FEV1 reached ≥ 70% predicted, the subject continued to receive the following standard treatment and assessment during the study treatment period:
  * Assessment of subject's signs and symptoms
  * Completion of a dyspnea index scale
  * Supplemental oxygen to maintain oxygen saturation, as measured by pulse oximetry of ≥ 90%
  * Albuterol (2.5 mg) via nebulizer given hourly NOTE: Albuterol (2.5 mg) via nebulizer and/or Ipratropium (0.5 mg) via nebulizer may have been given up to every 20 minutes and every hour, respectively, if deemed to be indicated by the Investigator.
  * Spirometry completed within 10 minutes of nebulizer treatments, followed by
  * Reassessment of signs and symptoms. If the subj
- MN-221 Placebo i.v. Infusion: MN-221 Placebo i.v. infusion. Until the subject's FEV1 reached ≥ 70% predicted, the subject continued to receive the following standard treatment and assessment during the study treatment period: Assessment of subject's signs and symptoms,Completion of a dyspnea index scale,Supplemental oxygen to maintain oxygen saturation, as measured by pulse oximetry of ≥ 90%,Albuterol (2.5 mg) via nebulizer given hourly. NOTE: Albuterol (2.5 mg) via nebulizer may have been given up to every 20 minutes if deemed to be indicated by the Investigator.
  * Ipratropium (0.5 mg) via nebulizer may have been given every hour if deemed to be indicated by the Investigator.
  * Spirometry completed within 10 minutes of nebulizer treatments, followed by
  * Reassessment of signs and symptoms. If the subject did not improve to FEV1 ≥70% of predicted during the study treatment period, the subject may have continued to receive further treatment, including hospital admission, at the discretion of the Investigator.
- 1,000-1,080 μg MN-221 i.v.: 16 μg/minute for 15 minutes followed by 8 μg/minute for 105 minutes (total dose of 1,080 μg). Among the subjects in the 1,000 - 1,080 μg group, per protocol instructions, the two subjects originally randomized to receive 1,080 μg MN-221 were infused with study drug over a 120-minute period and the 1 subject originally randomized to receive 450 μg who actually received 1,000 μg was infused with study drug over a 15-minute period. Although there was this difference in infusion time, it was deemed appropriate to group these 3 subjects in the same dose group.
- 450 μg MN-221 i.v. for 15 Minutes: 30 μg/minute for 15 minutes (total dose of 450 μg) administered i.v.
- 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes: Two subjects were randomized to receive 450 μg dose i.v. Instead, Subject 0010015 received 1,995 μg i.v. over 15 minutes infusion; Subject 0010016 received 1,995 μg i.v. over 25 minutes infusion.
Period: Overall Study
Arm/Group | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes | MN-221 Placebo i.v. Infusion | 1,000-1,080 μg MN-221 i.v. | 450 μg MN-221 i.v. for 15 Minutes | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes
Started | 5 | 13 | 3 | 6 | 2
Completed | 5 | 12 | 3 | 6 | 2
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes | MN-221 Placebo i.v. Infusion | 1,000-1,080 μg MN-221 i.v. | 450 μg MN-221 i.v. for 15 Minutes | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes | Total
Number analyzed (Participants) | 5 | 13 | 3 | 6 | 2 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 3 | 6 | 2 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.2 (11.56) | 42.6 (9.7) | 22.3 (3.21) | 39.2 (9.77) | 45 (0.0) | 37.83 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 3 | 6 | 2 | 21
  Male | 2 | 6 | 0 | 0 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 13 | 3 | 6 | 2 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change of FEV1 (Forced Expiratory Volume in 1 Second) Expressed as Percent of Predicted After Two Doses of Albuterol (5 mg Each) and Ipratropium (0.5 mg Each) When Compared to FEV1 at Hour 2 After the Start of the Infusion of MN-221 or Placebo.
Description: The primary efficacy summary was change from Baseline in FEV1 (percent predicted), at Hour 2. Baseline was defined as FEV1 (percent predicted) after two doses of albuterol (5 mg each) and ipratropium (0.5 mg each) and FEV1 (percent predicted) FEV1 at Hour 2 was defined as the FEV1 (percent predicted) at 2 hours after the start of the infusion of MN-221 or placebo. Change from Baseline in FEV1 (percent predicted), was summarized by treatment group at Hour 2.
Time Frame: Baseline and Hour 2
Population: The analysis was performed on the Intention-to-Treat (ITT) population. Twenty-nine subjects met the study entry criteria, provided written informed consent, and were enrolled in the study.
Measure: Mean (Full Range); unit: FEV1 (percent of predicted)
Arm/Group | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes | MN-221 Placebo i.v. Infusion | 1,000-1,080 μg MN-221 i.v. | 450 μg MN-221 i.v. for 15 Minutes | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes
Number analyzed (Participants) | 5 | 13 | 3 | 6 | 2
FEV1 (percent of predicted) | 16.57 (11.17) [4.8 to 44.7] | 3.88 (7.79) [-13.2 to 19.9] | 3.03 [-0.4 to 6.0] | 4.27 [-3.3 to 11.9] | -0.82 [-2.4 to 0.8]

2. Secondary Outcome: FEV1 (L) The Forced Expiratory Volume in One Second as Measured in Liters Per Second.
Description: FEV1 (L) was determined over time using a spirometer. Measure the mean change in FEV1 (L) from Baseline.
Time Frame: Baseline to Hour 2
Population: 29 subjects experiencing an acute exacerbation of asthma were at approximately 8 ED sites. The sample size was based on feasibility and precedent for this type of study, rather than statistical considerations.
Measure: Mean (Full Range); unit: liters per second
Groups:
- MN-221 at 16.0 μg/Min for 15 Min (Total 240 μg): The dosing scheme that consisted of a 15-minute infusion was based on PK (pharmacokinetic) modeling performed using data from the previous MN-221 studies that enrolled either healthy volunteers or subjects with stable mild to moderate asthma.
- Placebo Administered Intravenously: Initial dose group received MN-221 placebo intravenously for 15 minutes. For a subsequent dose group that was scheduled for a longer intravenous infusion of the study drug, subjects received MN-221 placebo intravenously for 15 minutes followed by MN-221 intravenously for 105 minutes.
- 450 μg MN-221 Given i.v.: The Data Safety Monitoring Board convened and recommended that the next highest scheduled can be administered to subjects. They received MN-221 at 30 μg/minute for 15 minutes (total dose 450 μg).
- 1,000-1,080 μg MN-221 Given i.v. for 15 Minutes: The Data Safety Monitoring Board recommended that subjects can receive MN-221 at 16 μg/minute for 15 minutes followed by 8 μg/minute for 105 minutes (total dose 1000-1080 μg).
- 1,995 MN-221 Administered i.v. for 15 Minutes and 25 Minutes: One subject that was randomized to receive 450 MN-221 intravenously for 15 minutes was administered 1995 micrograms. Another subject that was randomized to receive 450 micrograms for 15 minutes actually received a dose of 1995 micrograms MN-221 intravenously for 25 minutes.
Arm/Group | MN-221 at 16.0 μg/Min for 15 Min (Total 240 μg) | Placebo Administered Intravenously | 450 μg MN-221 Given i.v. | 1,000-1,080 μg MN-221 Given i.v. for 15 Minutes | 1,995 MN-221 Administered i.v. for 15 Minutes and 25 Minutes
Number analyzed (Participants) | 5 | 13 | 6 | 3 | 2
liters per second | 0.60 [0.14 to 1.67] | 0.10 [-0.51 to 0.54] | 0.12 [-0.09 to 0.33] | 0.10 [-0.02 to 0.22] | -0.02 [-0.07 to 0.02]

3. Secondary Outcome: Hospital Admission Rate During Visit 1
Description: After a patient in the emergency department (ED) presents with an acute exacerbation of asthma, the hospital proceeds with SOC procedures for this condition. Despite treatment in the ED, it is sometimes necessary to admit the patient into the hospital. In the study described here, the rate of hospital admissions was recorded.
Time Frame: Hour -1.5 through Hour 5
Measure: Number; unit: participants
Arm/Group | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes | MN-221 Placebo i.v. Infusion | 1,000-1,080 μg MN-221 i.v. | 450 μg MN-221 i.v. for 15 Minutes | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes
Number analyzed (Participants) | 5 | 13 | 3 | 6 | 2
participants | 0 | 7 | 0 | 3 | 1

ADVERSE EVENTS:
Arm/Group | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes | MN-221 Placebo i.v. Infusion | 1,000-1,080 μg MN-221 i.v. | 450 μg MN-221 i.v. for 15 Minutes | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes
Serious Adverse Events (participants affected / at risk) | 0/5 | 4/13 | 0/3 | 1/6 | 1/2
Other Adverse Events (participants affected / at risk) | 3/5 | 6/13 | 0/3 | 1/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes (N=5) | MN-221 Placebo i.v. Infusion (N=13) | 1,000-1,080 μg MN-221 i.v. (N=3) | 450 μg MN-221 i.v. for 15 Minutes (N=6) | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes (N=2)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Laboratory results were significant for elevated white blood cell count of 28,000 cells/microliter.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240 μg MN-221 i.v. (Intravenous) Infusion for 15 Minutes (N=5) | MN-221 Placebo i.v. Infusion (N=13) | 1,000-1,080 μg MN-221 i.v. (N=3) | 450 μg MN-221 i.v. for 15 Minutes (N=6) | 1,995 μg MN-221 i.v. Over 15 Minutes and 25 Minutes (N=2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (19) | 6 (12) | 0 (0) | 1 (3) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monocyte count decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less